CLINICAL TRIAL: NCT00750919
Title: A Twenty-six Weeks, Open-label Extension Trial to Evaluate Safety and Efficacy of Org 50081 (Esmirtazapine) in Outpatients With Chronic Primary Insomnia Who Completed Clinical Trial Protocol 21106
Brief Title: Twenty-six Week Extension Trial of Org 50081 (Esmirtazapine) in Outpatients With Chronic Primary Insomnia (176003/P05721/MK-8265-007)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This trial was stopped prematurely due to the Sponsor's decision not to continue the development of esmertazapine for this indication.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05721; 176003 (Other: Organon Protocol Number); 2007-005237-10 (EudraCT Number)
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Results first posted 2014-06-24 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Sleep Initiation and Maintenance Disorders; Mental Disorders; Dyssomnias; Sleep Disorders; Sleep Disorders, Intrinsic
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Mental Disorders; Dyssomnias; Sleep Wake Disorders; Sleep Disorders, Intrinsic | interventions — Mirtazapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Esmirtazapine (Experimental): Participants receive esmirtazapine 4.5 mg tablet, orally, once daily (QD) for up to 6 months.
  Interventions: Drug: esmirtazapine

INTERVENTIONS:
Drug: esmirtazapine

SUMMARY:
This trial is a 26-week, open label extension trial to investigate safety and explore efficacy of esmertazapine in participants with insomnia who completed protocol 21106/P05701/MK-8265-002 (NCT00631657).

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent
* Completed clinical trial 21106/P05701/MK-8265-002

Exclusion Criteria:

* Any (serious) adverse event, medical condition or required concomitant medication deemed relevant for exclusion in trial 21106/P05071/MK-8265-002 as judged by the investigator
* Were significantly non compliant with protocol criteria and procedures of trial 21106/P05701/MK-8265-002, as judged by the investigator
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2008-10-07 (Actual); Primary Completion 2010-03-10 (Actual); Study Completion 2010-03-10 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Ivgy-May N, Hajak G, van Osta G, Braat S, Chang Q, Roth T. Efficacy and safety of esmirtazapine in adult outpatients with chronic primary insomnia: a randomized, double-blind placebo-controlled study and open-label extension. J Clin Sleep Med. 2020 Sep 15;16(9):1455-1467. doi: 10.5664/jcsm.8526. PMID 32351205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed P05701 (Base study NCT00631657) were eligible to enroll on P05721 (Extension study).
Period: Overall Study
Arm/Group | Esmirtazapine
Started | 184
Completed | 126
Not Completed | 58
Not completed — Adverse Event | 9
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 8
Not completed — Could not cooperate, unrelated to trial | 4
Not completed — Other | 36

BASELINE CHARACTERISTICS:
Arm/Group | Esmirtazapine
Number analyzed (Participants) | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111
  Male | 73

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Sleep Time (TST)
Description: TST was defined as the time recorded for sleep diary question 6 "how much time did you actually spend sleeping" as reported by the participants using a LogPad (hand-held electronic data capture device). Baseline was defined as the TST from the last week of the base study. Daily diary data were converted to weekly averages. For each treatment week the non-missing diary data of that week were taken into account; if a treatment week had three non-missing morning diaries or less, the data of the previous week were taken into account, weighing the data of both weeks, using the number of observed diaries as weights (weighted mean); if no diary data were available for a treatment week the data were considered as missing and were not imputed.
Time Frame: Baseline and Week 26
Population: The All-Subjects-Treated (AST) population consisted of all participants who received at least one dose of esmertazapine in the extension study.
Measure: Mean (Standard Deviation); unit: Minutes per night
Arm/Group | Esmirtazapine
Number analyzed (Participants) | 184
Minutes per night
  Baseline measure (n=184) | 368.1 (91.5)
  Change from baseline at Week 26 (n=123) | 9.7 (56.1)

2. Secondary Outcome: Change From Baseline in Sleep Latency (SL)
Description: SL was defined as the time recorded for sleep diary question 3 "how long did it take you to fall asleep', " as reported by the participants using a LogPad (hand-held electronic data capture device). Baseline was defined as the SL from the last week of the base study. Daily diary data were converted to weekly averages. For each treatment week the non-missing diary data of that week were taken into account; if a treatment week had three non-missing morning diaries or less, the data of the previous week were taken into account, weighing the data of both weeks, using the number of observed diaries as weights (weighted mean); if no diary data were available for a treatment week the data were considered as missing and were not imputed.
Time Frame: Baseline and Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes per night
Arm/Group | Esmirtazapine
Number analyzed (Participants) | 148
Minutes per night
  Baseline measure (n=184) | 38.7 (32.0)
  Change from baseline at Week 26 (n=123) | -1.5 (39.1)

3. Secondary Outcome: Change From Baseline in Wake Time After Sleep Onset (WASO)
Description: WASO was defined as the time recorded for sleep diary question 5 "how much time were you awake, after falling asleep initially" as reported by the participants using a LogPad (hand-held electronic data capture device). Baseline was defined as the WASO from the last week of the base study. Daily diary data were converted to weekly averages. For each treatment week the non-missing diary data of that week were taken into account; if a treatment week had three non-missing morning diaries or less, the data of the previous week were taken into account, weighing the data of both weeks, using the number of observed diaries as weights (weighted mean); if no diary data were available for a treatment week the data were considered as missing and were not imputed.
Time Frame: Baseline and Week 26
Population: The AST population consisted of all participants who received at least one dose of esmertazapine in the extension study.
Measure: Mean (Standard Deviation); unit: Minutes per night
Arm/Group | Esmirtazapine
Number analyzed (Participants) | 148
Minutes per night
  Baseline measure (n=184) | 40.0 (43.5)
  Change from baseline at Week 26 (n=123) | -5.4 (32.3)

4. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An adverse event is any unfavorable and unintended change in the structure, function, or chemistry of the body whether or not considered related to the study treatment.
Time Frame: Up to 30 weeks
Population: The AST population consisted of all participants who received at least one dose of esmertazapine in the extension study.
Measure: Number; unit: Participants
Arm/Group | Esmirtazapine
Number analyzed (Participants) | 184
Participants | 127

5. Primary Outcome: Number of Participants Discontinuing Due to AEs
Description: as for outcome 4
Time Frame: Up to 26 weeks
Population: The AST population consisted of all participants who received at least one dose of esmertazapine in the extension study.
Measure: Number; unit: Participants
Arm/Group | Esmirtazapine
Number analyzed (Participants) | 184
Participants | 9

ADVERSE EVENTS:
Time Frame: Nonserious AEs were collected from first dispensing of study drug up to 7 days after last dose of study drug. Serious AEs were collected from first dispensing of study drug up to 30 days after last dose of study drug.
Arm/Group | Esmirtazapine
Serious Adverse Events (participants affected / at risk) | 3/184
Other Adverse Events (participants affected / at risk) | 59/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esmirtazapine (N=184)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Strabismus correction (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esmirtazapine (N=184)
Nasopharyngitis (Infections and infestations) | 19 (20)
Weight increased (Investigations) | 11 (12)
Headache (Nervous system disorders) | 10 (13)
Somnolence (Nervous system disorders) | 10 (11)
Insomnia (Psychiatric disorders) | 23 (23)

LIMITATIONS AND CAVEATS:
This study was terminated due to the Sponsor's decision not to continue development of esmertazapine for this indication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less